CLINICAL TRIAL: NCT02448017
Title: Effects of Herbst Appliance Therapy to Improve Airway Dimension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HKCTR-1858
Record Dates: First submitted 2015-02-04; First posted 2015-05-19 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Angle Class II
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- The Herbst appliance (Active Comparator): Orthodontic functional appliance
  Interventions: Device: The Herbst appliance
- Twin block appliance (Active Comparator): Orthodontic functional appliance
  Interventions: Device: Twin block appliance

INTERVENTIONS:
Device: The Herbst appliance — Orthodontic functional appliance
  Arms: The Herbst appliance
Device: Twin block appliance — Orthodontic functional appliance
  Arms: Twin block appliance

SUMMARY:
Herbst appliance is one of the most popular fixed functional appliances to treat orthodontic patients with small lower jaws. Since small lower jaws are reported to be one of the main reasons to induce sleep disordered breathing(SDB) of children, Herbst appliance can be used to treat SDB children. Previously no study compared the effects of Herbst appliance therapy with removable functional appliance on airway dimension, so it still remains unclear which kinds of functional appliance is more suitable for improving airway dimension. This study will assess the effect of Herbst appliance on airway dimension and compare the effects with those of twin block appliance (a popular 24 hours used removable functional appliance, and also commonly used to treat adult sleep apnea).

DETAILED DESCRIPTION:
Sleep disordered breathing (SDB) is an important paediatric problem. It is estimated that 3.2% to 12.1% of children have habitual snoring and 0.7% to 10.3% have obstructive sleep apnea syndrome (OSAS). Children OSAS is associated with a series of daytime and nighttime signs and symptoms. Nighttime symptoms include heavy snoring, restless sleep, heavy seating and enuresis, etc. Daytime symptoms include excessive daytime sleepiness and abnormal behavior such as aggressiveness and hyperactivity, etc. Untreated OSAS was reported to result in serious morbidity, such as failure to thrive, poor learning, attention deficit and hyperactivity disorder, etc.

There is an increasing concern related to sleep disordered breathing(SDB) of children by orthodontists. Since not only the tonsilar and adenoid hypertrophy is the main cause of paediatric OSA, but also craniofacial anomalies such as retrognathic mandible, narrow maxillary palatal arch and increased lower facial height can also contribute to it, orthopedic treatment such as rapid maxillary expansion (RME) and mandibular advancement device (MAD) may potentially permanently cure the children OSA. RME which is used to widen maxilla, thus increasing the nasal cavity and improving the nasal flow, has been thoroughly researched. However, only a few previous studies focused on the treatment effect of MAD for treating OSA children. These studies showed sorts of MAD such as jaw-positioning appliance, mono-block, and Herbst appliance were effective to OSA children, but it remains unclear how to choose a functional appliance, and if there is any treatment difference between removable functional appliance and fixed functional appliance for improving airway dimension.

ELIGIBILITY:
Inclusion Criteria:

1. Class II malocclusion

Exclusion Criteria:

1. Cleft lip and palate
2. Craniofacial syndrome

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2012-07; Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
The cephalometric measurement of dimensional change of upper way following 2-phase orthodontic treatment | 3 years two-phase treatment with functional appliance and fixed appliance
  The two-phase treatment effects of Herbst and twin-block appliances on the upper airway are to be compared based on the lateral cephalometric analysis at three time points (T0: pre-treatment; T1: following 1 year functional appliance treatment; T3: following 2 years fixed appliance treatment). The parameters of lateral cephalometric analysis include the measurements of the depth of pharynx, the size of soft palate and the position of the hyoid bone.

SECONDARY OUTCOMES:
The three-dimensional change of upper way following 2-phase orthodontic treatment in magnetic resonance images | 3 years two-phase treatment with functional appliance and fixed appliance
  The two-phase treatment effects of Herbst and twin-block appliances on the upper airway are to be compared based on the analyses of magnetic resonance images at three time points (T0: pre-treatment; T1: following 1 year functional appliance treatment; T3: following 2 years fixed appliance treatment).The analyses include measurements of the depth and width of pharynx, the size of soft palate and the tongue.

CONTACTS AND LOCATIONS:
Overall Officials: Yanqi Yang, Principal Investigator — The Paediatric dentistry and orthodontic department, Faculty of Dentistry, the University of Hong Kong
Locations (1):
- Faculty of Dentistry, the University of Hong Kong, Hong Kong, Hong Kong, China